CLINICAL TRIAL: NCT00944242
Title: Bioequivalence Study of Sertraline 100 mg Tablet and ZOLOFT Following a 100 mg Dose in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: 40485
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline
Drug: Sertraline Hydrochloride

SUMMARY:
* Objective:

  * To compare the rate and extent of absorption of Torrent Pharmaceuticals Limited, India, sertraline and Pfizer, Inc., USA (Zoloft) sertraline, administered as a 1X100 mg tablet, under fasted conditions.
* Study Design:

  * Single-dose, open-label, randomized two-way crossover.

ELIGIBILITY:
* Inclusion Criteria:

  * Male or female, smoker or non smoker, 18 years of age and older.
  * Capable of consent.
  * BMI>= 19.0 and <30.0 kg/m2
* Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illness or surgery within 4 weeks prior to the administration of the study medication.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities or vital sign abnormalities(blood pressure).
* History of significant alcohol or drug abuse within one year prior to the screening visit.
* History or allergic reactions to heparin, sertraline or other related drugs.
* Use of an investigational drug or participation in an investigational study with in 30 days prior to administration of the study medication.
* Clinically significant history of gastrointestinal pathology, liver or kidney disease, neurological, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* History of seizures, suicide attempt, bipolar disorder or manic episodes.
* Depot injection or an implant of any drugs with in 6 months prior to administration of study medication.
* Breastfeeding subject.
* Positive urine pregnancy test at screening.
* female subject of child bearing potential having unprotected sexual intercourse with any non-sterile mail partner within 14 days prior to study drug administration.

Acceptable methods of contraception:

1. Intra-uterine contraceptive device(placed at least 4 weeks prior to study drug administration)
2. Condom or diaphragm + spermicide.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anapharm Inc., Montreal, Quebec, Canada